CLINICAL TRIAL: NCT05747326
Title: A Doublelet Metronomic Chemotherapeutic Regimen With Oral Vinorelbine and Capecitabine in Advanced HER2-negative Breast Cancer Patients: A Monocentric Retrospective Study in China
Brief Title: Oral Vinorelbine and Capecitabine in Advanced HER2-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: m-VCAP1
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; metronomic treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Intervention Model Description: This study was a prospective, single-arm, open-label phase II clinical trial conducted at National cancer center in China. The eligible patients were enrolled to receive oral metronomic vinorelbine 40 mg on day 1, day 3, day 5 every week (Monday, Wednesday, and Friday) and capecitabine 500mg three times daily (tid) after meals every 3 weeks. Until disease progression or unacceptable toxicity occurred, or the patient refused medication, vinorelbine and capecitabine were administered continuously without drug-free periods over 21-day cycles.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The eligible patients were enrolled to receive oral metronomic vinorelbine 40 mg on day 1, day 3, day 5 every week (Monday, Wednesday, and Friday) and capecitabine 500mg three times daily (tid) after meals every 3 weeks. Until disease progression or unacceptable toxicity occurred, or the patient refused medication, vinorelbine and capecitabine were administered continuously without drug-free periods over 21-day cycles.
  Interventions: Drug: oral vinorelbine and capecitabine

INTERVENTIONS:
Drug: oral vinorelbine and capecitabine — The eligible patients were enrolled to receive oral metronomic vinorelbine 40 mg on day 1, day 3, day 5 every week (Monday, Wednesday, and Friday) and capecitabine 500mg three times daily (tid) after meals every 3 weeks. Until disease progression or unacceptable toxicity occurred, or the patient refused medication, vinorelbine and capecitabine were administered continuously without drug-free periods over 21-day cycles.
  Other Names: metronomic agents (vinorelbine and capecitabine )

SUMMARY:
This study was a prospective, single-arm, open-label phase II clinical trial conducted at National cancer center in China.

DETAILED DESCRIPTION:
Metronomic chemotherapy is a relatively low-dose, high-frequency, continuous application of cytotoxic agents. Phase I/II VICTOR-1 studies have shown that the dual oral beat combination of vincristine and capecitabine is highly active and well tolerated in patients with locally advanced or metastatic breast cancer. The long-term efficacy of oral two-metronomic agents (vinorelbine and capecitabine) in Chinese advanced HER-2 negative breast cancer patients stays unclear. The current study was designed to explore the efficacy of oral two-metronomic agents (vinorelbine and capecitabine) in advanced HER-2 negative patient China.

ELIGIBILITY:
Inclusion Criteria:

* female;
* aged ≥ 18 years and ≤75 years;
* histologically proved metastatic HER-2 negative breast cancer. HER2-negative status determined by situ hybridization (FISH) or immunohistochemistry (IHC) (IHC 0, 1+, 2+ and/or FISH HER2 negative);
* at least one measurable or evaluable lesion based on RECIST 1.1 criteria;
* estimated life expectancy ≥ 3 months;
* normal heart, liver, and kidney function;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
* informed consent signed by the participants

Exclusion Criteria:

* received neoadjuvant or adjuvant therapy containing vinorelbine or capecitabine within one year prior to treatment initiation;
* participated in other new drug clinical trials within 4 weeks before enrollment;
* inflammatory breast cancer;
* symptomatic visceral disease;
* second primary malignancy;
* mental disorder.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | At 1 year
  1-year progression-free survival (PFS1). Evidence of local recurrence, distant metastasis, or death from any cause within 1 year counted as events in the time-to-event Kaplan-Meier analysis of progression-free survival. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions

SECONDARY OUTCOMES:
Proportion of Confirmed Response, Defined as a Partial Response (PR) or Better | Up to 1 year
  Confirmed response will be evaluated using all cycles. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR Confirmed response will be evaluated using all cycles. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Study Director — National Cancer Center/National Clinical Research Center for Cancer
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual anonymized participant data will not be shared.

REFERENCES:
- [Derived] Chai Y, Liu J, Jiang M, He M, Wang Z, Ma F, Wang J, Yuan P, Luo Y, Xu B, Li Q. A phase II study of a doublet metronomic chemotherapy regimen consisting of oral vinorelbine and capecitabine in Chinese women with HER2-negative metastatic breast cancer. Thorac Cancer. 2023 Aug;14(23):2259-2268. doi: 10.1111/1759-7714.15011. Epub 2023 Jul 4. PMID 37402471